CLINICAL TRIAL: NCT05202184
Title: Non Transplantable Recurrence After Percutaneous Thermal Ablation of ≤3cm HCC: Predictors and Implications for Treatment Allocation
Brief Title: Non Transplantable Recurrence After Percutaneous Thermal Ablation of HCC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0436_3
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: HCC
Keywords: With or without cirrhosis; BCLC0 or A; No extra-hepatic disease; Radiofrequency ablation; Microwave ablation; Liver transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Percutaneous thermal ablation of small HCC: Percutaneous thermal ablation of small HCC
  Interventions: Procedure: Percutaneous thermal ablation

INTERVENTIONS:
Procedure: Percutaneous thermal ablation — All thermoablation procedures were performed percutaneously under ultrasound and/or CT guidance

SUMMARY:
Percutaneous thermal ablation (PTA), resection and liver transplantation (LT) are the standard curative options for hepatocellular carcinoma (HCC). LT yields the best long-term outcomes but is limited by graft shortage. Thus, patients with ≤3cm HCC are mainly treated by PTA although recurrence is frequent and may occur outside transplant criteria. However, data on non transplantable recurrence (NTR) following PTA are lacking. Therefore, the investigators investigated the incidence and predictors of NTR among transplantable patients with ≤3cm HCC(s) treated by PTA, in order to stratify them according to their NTR risk and to improve treatment allocation.

DETAILED DESCRIPTION:
Consecutive patients undergoing PTA for HCC between January 2015 and December 2020 were included. Data were collected from our prospective database. This study was approved by our institutional review board (NCT03428321 [www.clinicaltrials.gov]) and written informed consent was obtained from all patients. Inclusion criteria were: HCC diagnosed by histopathology or by EASL imaging criteria, HCC ≤30mm, 1 - 3 tumor nodules, follow-up<3 months, no prior or combined treatment with intra-arterial therapy, potentially transplantable patient (ie, ≤70yr, AFP-score≤2 (7), no macroscopic portal vein invasion or extra-hepatic metastasis, no major comorbidity precluding LT).

Patient's and liver's characteristics were collected including: age, sex, HCC-naïve status, body mass index (BMI), diabetes mellitus, liver steatosis, cirrhosis, cause for hepatopathy, AFP serum level, Child-Pugh, MELD and Albumin-Bilirubin (ALBI) scores and preablative biological data.

Occurrence of NTR after PTA will be analyzed in a competing risks framework, with transplantation and death as competing events. Covariates associated with NTR were analyzed using Fine-Gray proportional sub-distribution hazards models.

Recurrence-free survival (RFS) will be defined as the time from PTA until the first recurrence, death, or last follow-up. OS will be defined as the interval between PTA and death (any cause) or last follow-up. Survival curves will be estimated using the Kaplan-Meier method and compared with the log-rank test.

ELIGIBILITY:
Inclusion criteria :

* HCC diagnosed by histopathology or by EASL imaging criteria
* HCC ≤30mm, 1 - 3 tumor nodules, follow-up<3 months
* no prior or combined treatment with intra-arterial therapy
* potentially transplantable patient (ie, ≤70yr, AFP-score≤2 (7), no macroscopic portal vein invasion or extra-hepatic metastasis, no major comorbidity precluding LT).

Exclusion criteria:

- age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing PTA for HCC between January 2015 and December 2020 were included. Data were collected from our prospective database at the Department of Radiology St-Eloi University Hospital - Montpellier School of Medicine France.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of non transplantable recurrence | 1 day
  Incidence of non transplantable recurrence

CONTACTS AND LOCATIONS:
Overall Officials: BORIS GUIU, PU-PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC